CLINICAL TRIAL: NCT07005973
Title: Effects of Mobile-based Mindfulness Intervention to Reduce Preoperative Anxiety for Patients Undergoing Elective Surgery: A Pilot Randomized Controlled Trial
Brief Title: Effects of Mobile-based Mindfulness Intervention to Reduce Preoperative Anxiety for Patients Undergoing Elective Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, KWAN KIT HANG, Advanced Practice Nurse, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB-2025-146-3
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Mobile-based Mindfulness Intervention to Reduce Preoperative Anxiety; Pre-operative Anxiety; Postoperative Pain; Postoperative Use of Analgesics
Keywords: Mobile-based mindfulness; pre-operative anxiety; post-operative pain; postoperative use of analgesics
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients will receive usual care from surgeon, anesthetist and perioperative team including the delivery of operation related information, environment of operating theatre, the process of anesthesia, postoperative care from recovery room to discharge, etc.
- Intervention group (Experimental): Patients will be provided with usual care by surgeon, anesthetist and perioperative team, and they will be asked to install a validated mindfulness based mobile app during the PAS session. Orientation and teaching on the use of the mobile app will be carried out by research team. Return demonstration by patients will be performed at the end to ensure they are capable to use the app at home independently.
  Interventions: Behavioral: mobile-based mindfulness intervention

INTERVENTIONS:
Behavioral: mobile-based mindfulness intervention — Patients will be provided with usual care by surgeon, anesthetist and perioperative team, and they will be asked to install a validated mindfulness based mobile app during the PAS session. Orientation and teaching on the use of the mobile app will be carried out by research team. Return demonstration by patients will be performed at the end to ensure they are capable to use the app at home independently.
  A minimum of 4-week intervention duration with session lengths of 1 min, 3 days per week is set for this study.
  Patients will be distributed a dairy log to record the frequency and duration of mindfulness practice and submit to the researcher on the day of admission. Follow up on patient's progress through phone call or whatsapp will be provided by the researcher to ensure patient's adherence to the intervention on a bi-weekly basis.
  Arms: Intervention group

SUMMARY:
This study is a pilot randomized controlled trial (RCT) conducted at Tin Shui Wai Hospital to evaluate the effectiveness of a mobile-based mindfulness intervention in reducing preoperative anxiety among patients scheduled for elective surgery.

Aim: To determine if a 4-week mindfulness program delivered via a mobile app can reduce preoperative anxiety, compared to standard care.

Design:

Parallel-arm RCT with 40 participants (20 in each group). Participants are randomly assigned to either the intervention group (mobile-based mindfulness intervention + usual care) or control group (usual care only).

The intervention uses a free and anonymous mindfulness mobile app developed by The University of Hong Kong.

Primary Outcome:

Preoperative anxiety level on the day of surgery, will be assessed using the STAI-S questionnaire.

Secondary Outcomes:

Postoperative pain levels, use of analgesics, emergency department revisit rate, and user satisfaction with the app.

Data Collection:

Anxiety levels are measured at baseline and before surgery. Pain levels and analgesic use are recorded postoperatively. Emergency visits and usability feedback are collected post-discharge.

Significance:

The study addresses a gap in evidence for mobile mindfulness interventions in Chinese surgical patients.

Findings may support the integration of low-cost, app-based mindfulness into preoperative care.

DETAILED DESCRIPTION:
Preoperative anxiety is a common phenomenon being reported in 60-80% of patients who are undergoing a surgical procedure and it was shown to be associated with negative postoperative outcomes such as suboptimal pain control, sleep disturbances, delayed wound healing, prolonged length of hospitalization and dissatisfying patients' hospitalization experience as a result. The current practice being adopted to minimize the level of anxiety in preoperative patients includes pharmacological and non-pharmacological approach. Pharmacological interventions include sedative and anti-anxiety drugs can be used before an operation to improve patient's emotion, however, studies have shown that adverse reactions on respiratory and central nervous system may be encountered, leading to a negative outcome of the operation. On the other hand, non-pharmacological interventions such as spiritual support, hypnosis, acupuncture, interview, cognitive behaviour therapy (CBT) and meditation are shown to be an effective strategy to alleviate the preoperative anxiety by anesthesiologists.

Mindfulness is a meditation concept originally introduced from India and has been developed into a structured approach for stress reduction treatment, nowadays commonly being adapted in both clinical and non-clinical setting. Mindfulness-based interventions (MBIs) have demonstrated efficacy in improving various clinical outcomes especially in reducing stress and anxiety. Mindfulness-based stress reduction (MBSR) program is a well-known MBI widely being used in various clinical conditions include the management on chronic pain, cancer, vascular disease and preoperative anxiety. However, traditional MBIs programs are extensive and required face-to-face training conducted by a well-trained qualified instructor. The standard MBSR program is intensive, consists of a 2.5 hours weekly group-based face-to-face classes lasting for 8 weeks plus a one full day retreat at the end of the program. Taking into consideration of the long duration and a certified instructor are required for the standard MBSR training program, delivery of mobile-based mindfulness interventions via the mobile app was introduced as an alternative platform to practice mindfulness making it feasible, accessible, acceptable and inexpensive in reducing psychological distress.

According to the systematic review, positive impact of mobile-based mindfulness interventions with the enhancement on mental health treatment was found and mobile-based mindfulness interventions were also found to be promising as an adjunct intervention only to improve mindfulness skills and depressive symptoms. In view of the inconsistency of clinical outcomes on mobile-based mindfulness interventions among systematic reviews, a randomized controlled trial to examine the effectiveness of mobile-based mindfulness interventions for reduction of preoperative anxiety need to be studied in local context. Furthermore, the effects of mobile-based mindfulness interventions on preoperative anxiety have been understudied in Chinese population and the recent systematic review has not identified in any Chinese study.

The aim of study is to examine the effects of mobile-based mindfulness intervention to reduce preoperative anxiety for patients undergoing elective surgery. We hypothesize that compared to standard care group, delivery of mobile-based mindfulness intervention can reduce preoperative anxiety for patients undergoing elective surgery.

A parallel-arm (mobile-based mindfulness intervention vs. usual care [active control]) randomized controlled trial (RCT) will be adapted in this study as RCT is the best study design to control for confounders.

This RCT study will be conducted in Tin Shui Wai Hospital. Approval and endorsement have been granted from Chief of Service (COS) of surgery department. The research proposal will be submitted to Hospital Authority Central Institutional Review Board (IRB) for ethical approval, and then it will be pre-registered in research registry at clinicaltrials.gov.

Patients with evidence of anxiety and meeting the inclusion criteria will be recruited to the trial directly during they attend the Pre-anaesthesia Assessment Service (PAS) in day ward of Tin Shui Wai Hospital.

Level of anxiety will be assessed through the State-Trait Anxiety Inventory Form Y (STAI-Y) which is divided into the measurement of state and trait anxiety. The original STAI was developed in 1970 and has been translated to more than 30 languages for cross-cultural research and clinical practice. STAI-Y has been proven that it is an appropriate and adequate instrument for anxiety related study in both research and clinical settings in accordance to various reliability and validity tests.

The STAI-Y is a 4-point Likert self-reported scale consisting of a total of 40 items, which are divided into two subscales: trait anxiety (STAI-T) and state anxiety (STAI-S), each containing 20 items. STAI-T is used to determine a person's underlying personality anxiety level as trait anxiety is a more stable tendency to react to stress with anxiety which reflecting the underlying part of a person's personality; while STAI-S is used to determine a person's current anxiety level as state anxiety is a temporary emotional state involving feelings of tension that can fluctuate in intensity and usually appears in preoperative patients. The STAI-All items are followed by a 4-point scale rating the frequency of feelings from "not at all" to "very much", and scoring from 1 to 4 each. The subtotal score ranged from 20 to 80 with higher scores indicated higher level of anxiety. A cut-off point of 39-40 has been suggested for detection of clinically relevant symptoms for the state anxiety scale. A validated Chinese version of STAI-Y questionnaire will be adapted in this study.

Patients' anxiety level will be assessed at 2 different time-points: baseline assessment will be conducted on the day of patients attending PAS clinic (T0); post treatment assessment on the day of admission before patients being sent to operation theater (T1).

All patients attend the PAS clinic will be initially distributed the STAI-T questionnaire to fill in to detect subjects with potential underlying anxiety. A cutoff score of 40 is commonly used to define probable clinical levels of anxiety, therefore, patients with score 40 or above showed in questionnaire of STAI-T will be invited to participate in this clinical trial.

Research investigator will explain the details of the trial and answer all the questions raised by patients. These patients are then presented with the written information of the trial. Each participant will receive a written informed consent. As all patients' participation are on voluntary basis, they could withdraw from the study at any time without penalty during the trial.

Patients will be randomly allocated (1:1) into 2 groups: intervention group or control group.

For control group, patients will receive usual care from surgeon, anesthetist and perioperative team including the delivery of operation related information, environment of operating theatre, the process of anesthesia, postoperative care from recovery room to discharge, etc.

For intervention group, patients will be taught to exercise mindfulness on top of receiving usual care as control group. This group of patients will be helped to install a mobile app on mindfulness developed by the University of Hong Kong which is originally being used for the promotion of mental health among students and teachers in Hong Kong. The mobile app is now opened to the public and no pre-registration is required for using the app. The mobile app provides a platform with video and audio-guided soundtracks which includes body scan, mindful breathing, eating, stretching and natural sounds for public to practice mindfulness at home. Upon the recruitment, patients will be educated to use the app regularly at home until their scheduled surgery appointment. Interval phone follow up will be provided for the intervention group patients on the use of the mindfulness mobile app to ensure the compliance to the intervention and also to tackle with the difficulties they may encounter during the interventional period.

ELIGIBILITY:
Inclusion Criteria:

* adult (age>= 18 years old)
* scheduled to undergo non-emergency surgery under general anesthesia (GA)
* use of smart phone
* able to understand the Chinese language and express their feelings sufficiently
* STAI-T score >=40

Exclusion Criteria:

* unable to provide informed consent
* history or current treatment for psychological complaints
* serious physical or psychological co-morbidities
* hearing or vision impairment
* patients withdrawal from continuing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-operative anxiety level | From enrollment to the day of admission for surgery (at least 4 weeks)
  Pre-operative anxiety level on admission day of undergoing surgery: As mobile-based mindfulness intervention will be exercised by patients at home since last attendance to PAS session until the operation day (primary study endpoint). On the day of operation before patient being sent to the operation theatre (T1), patients will be asked to fill in the State-Trait Anxiety Inventory-State (STAI-S) questionnaire to document the level of anxiety. The score ranged from 20 to 80 with higher scores indicated higher level of anxiety.

SECONDARY OUTCOMES:
Postoperative pain level | From the day of admission to the day of discharge after surgery
  Patients undergoing surgery commonly experience pain after surgery and it may lead to a poor outcome. Study reported that 86% patients experienced pain after surgery and 75% had moderate to extreme pain during the immediate post-surgical period, with 74% still experienced pain after discharge. Mindfulness based intervention was also being reported to be an effective non-pharmacological technique in dealing with pain. Therefore, level of pain will be set as one of the secondary outcomes in this study. Pain intensity will be measured by a 11-point pain intensity numerical rating scale (PI-NRS), where 0=no pain and 10=worst possible pain given that PI-NRS is a widely used and validated instrument to measure clinical pain. Patients' pain level will be assessed before the surgery (T1); and immediately after surgery (T2).
Postoperative use of analgesics | From post-operation to the day of discharge
  In view of majority of patients experience pain after surgery, pain killer may be administrated during hospitalization. The frequency, choice of analgesics being used, dosage being given to patients for postoperative pain control will be retrieved and reviewed in the In-patient Medication Order Entry (IPMOE) record after patients discharged.
Number of times of revisiting emergency department after discharge | From the day of discharge to 1 month after surgery
  Limited studies have reported the relationship of the providence of anxiety reduction programme before surgery and the number of times of revisiting emergency department after discharge. Thus, number of times of revisiting emergency department due to post-operation related issues 1 month after discharge will be set as the secondary outcome to explore their correlation.
User Satisfaction | From enrollment to the day of discharge after surgery
  User satisfaction survey will be administered to the intervention group patients before they are being discharged so as to document their satisfaction level on using the mobile-based mindfulness intervention and to explore the feasibility of applying it in clinical setting in the future.

CONTACTS AND LOCATIONS:
Overall Officials: KIT HANG MR KWAN, Advanced Practice Nurse, Principal Investigator — Tin Shui Wai Hospital
Locations (1):
- Tin Shui Wai Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang R, Huang X, Wang Y, Akbari M. Non-pharmacologic Approaches in Preoperative Anxiety, a Comprehensive Review. Front Public Health. 2022 Apr 11;10:854673. doi: 10.3389/fpubh.2022.854673. eCollection 2022. PMID 35480569
- [Background] Zhang J, Gao Q. Validation of the trait anxiety scale for state-trait anxiety inventory in suicide victims and living controls of Chinese rural youths. Arch Suicide Res. 2012;16(1):85-94. doi: 10.1080/13811118.2012.641440. PMID 22289030
- [Background] Wong SH, Tan ZYA, Cheng LJ, Lau ST. Wearable technology-delivered lifestyle intervention amongst adults with overweight and obese: A systematic review and meta-regression. Int J Nurs Stud. 2022 Mar;127:104163. doi: 10.1016/j.ijnurstu.2021.104163. Epub 2021 Dec 18. PMID 35092872
- [Background] Spielberger, C.D., Gorsuch, R.C., Lushene, R.E. (1970). Manual for the State-Trait. Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Reynolds KA, Sommer JL, Roy R, Kornelsen J, Mackenzie CS, El-Gabalawy R. A Qualitative Analysis of the Impact of Preoperative Mindfulness-Based Stress Reduction on Total Knee Arthroplasty Surgical Experiences. Pain Manag Nurs. 2024 Aug;25(4):409-416. doi: 10.1016/j.pmn.2024.04.002. Epub 2024 May 2. PMID 38697887
- [Background] Plaza Garcia I, Sanchez CM, Espilez AS, Garcia-Magarino I, Guillen GA, Garcia-Campayo J. Development and initial evaluation of a mobile application to help with mindfulness training and practice. Int J Med Inform. 2017 Sep;105:59-67. doi: 10.1016/j.ijmedinf.2017.05.018. Epub 2017 May 31. PMID 28750912
- [Background] Maurice-Szamburski A, Auquier P, Viarre-Oreal V, Cuvillon P, Carles M, Ripart J, Honore S, Triglia T, Loundou A, Leone M, Bruder N; PremedX Study Investigators. Effect of sedative premedication on patient experience after general anesthesia: a randomized clinical trial. JAMA. 2015 Mar 3;313(9):916-25. doi: 10.1001/jama.2015.1108. PMID 25734733
- [Background] Marinelli V, Danzi OP, Mazzi MA, Secchettin E, Tuveri M, Bonamini D, Rimondini M, Salvia R, Bassi C, Del Piccolo L. PREPARE: PreoPerative Anxiety REduction. One-Year Feasibility RCT on a Brief Psychological Intervention for Pancreatic Cancer Patients Prior to Major Surgery. Front Psychol. 2020 Mar 5;11:362. doi: 10.3389/fpsyg.2020.00362. eCollection 2020. PMID 32194490
- [Background] Macrynikola N, Mir Z, Gopal T, Rodriguez E, Li S, Cox M, Yeh G, Torous J. The impact of mindfulness apps on psychological processes of change: a systematic review. Npj Ment Health Res. 2024 Mar 18;3(1):14. doi: 10.1038/s44184-023-00048-5. PMID 38609511
- [Background] Lu YJ, Lee MC, Chen CY, Liang SY, Li YP, Chen HM. Effect of Guided Imagery Meditation During Laparoscopic Cholecystectomy on Reducing Anxiety: A Randomized Controlled Trial. Pain Manag Nurs. 2022 Dec;23(6):885-892. doi: 10.1016/j.pmn.2022.07.003. Epub 2022 Jul 31. PMID 35922271
- [Background] Lonner, W.J., Ibrahim, F.A. (1989). Assessment in Cross-Cultural Counseling. Thousand Oaks, CA: Sage Publications Inc.
- [Background] Lin JY, Lu Y. Establishing a data monitoring committee for clinical trials. Shanghai Arch Psychiatry. 2014 Feb;26(1):54-6. doi: 10.3969/j.issn.1002-0829.2014.01.009. PMID 25114483
- [Background] Knowles KA, Olatunji BO. Specificity of trait anxiety in anxiety and depression: Meta-analysis of the State-Trait Anxiety Inventory. Clin Psychol Rev. 2020 Dec;82:101928. doi: 10.1016/j.cpr.2020.101928. Epub 2020 Oct 10. PMID 33091745
- [Background] Kain ZN, Sevarino F, Pincus S, Alexander GM, Wang SM, Ayoub C, Kosarussavadi B. Attenuation of the preoperative stress response with midazolam: effects on postoperative outcomes. Anesthesiology. 2000 Jul;93(1):141-7. doi: 10.1097/00000542-200007000-00024. PMID 10861157
- [Background] Julious, S. A. (2005). Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics : The Journal of the Pharmaceutical Industry, 4(4), 287-291.
- [Background] Jlala HA, French JL, Foxall GL, Hardman JG, Bedforth NM. Effect of preoperative multimedia information on perioperative anxiety in patients undergoing procedures under regional anaesthesia. Br J Anaesth. 2010 Mar;104(3):369-74. doi: 10.1093/bja/aeq002. Epub 2010 Feb 1. PMID 20124283
- [Background] In J. Introduction of a pilot study. Korean J Anesthesiol. 2017 Dec;70(6):601-605. doi: 10.4097/kjae.2017.70.6.601. Epub 2017 Nov 14. PMID 29225742
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Grutz K, Poch N. Meditation for Preoperative Anxiety and Postoperative Pain in Bariatric Surgery. J Perianesth Nurs. 2021 Oct;36(5):586-590. doi: 10.1016/j.jopan.2021.04.003. No abstract available. PMID 34688457
- [Background] Garland EL, Baker AK, Larsen P, Riquino MR, Priddy SE, Thomas E, Hanley AW, Galbraith P, Wanner N, Nakamura Y. Randomized Controlled Trial of Brief Mindfulness Training and Hypnotic Suggestion for Acute Pain Relief in the Hospital Setting. J Gen Intern Med. 2017 Oct;32(10):1106-1113. doi: 10.1007/s11606-017-4116-9. Epub 2017 Jul 12. PMID 28702870
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Emons WH, Habibovic M, Pedersen SS. Prevalence of anxiety in patients with an implantable cardioverter defibrillator: measurement equivalence of the HADS-A and the STAI-S. Qual Life Res. 2019 Nov;28(11):3107-3116. doi: 10.1007/s11136-019-02237-2. Epub 2019 Jun 22. PMID 31230167
- [Background] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Background] Creswell JD. Mindfulness Interventions. Annu Rev Psychol. 2017 Jan 3;68:491-516. doi: 10.1146/annurev-psych-042716-051139. Epub 2016 Sep 28. PMID 27687118
- [Background] Chen M, Huang Y, Zhang J, Wu Z, Lin C, Zheng B, Chen C, Li W. Impact of preoperative anxiety on postoperative outcomes in patients undergoing minimally invasive thoracoscopic surgery: A prospective cohort study. Eur J Surg Oncol. 2024 Oct;50(10):108605. doi: 10.1016/j.ejso.2024.108605. Epub 2024 Aug 13. PMID 39151308
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Beiranvand S, Noparast M, Eslamizade N, Saeedikia S. The effects of religion and spirituality on postoperative pain, hemodynamic functioning and anxiety after cesarean section. Acta Med Iran. 2014;52(12):909-15. PMID 25530054
- [Background] Ayers DC, Franklin PD, Trief PM, Ploutz-Snyder R, Freund D. Psychological attributes of preoperative total joint replacement patients: implications for optimal physical outcome. J Arthroplasty. 2004 Oct;19(7 Suppl 2):125-30. doi: 10.1016/j.arth.2004.06.019. PMID 15457431